CLINICAL TRIAL: NCT04516564
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose, First-In-Human Study Evaluating the Safety, Tolerability, and Pharmacokinetics of AK119 in Healthy Subjects
Brief Title: A Study of AK119 (Anti-CD73 Antibody), a Treatment for COVID-19, in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Akesobio Australia Pty Ltd (Industry)
Responsible Party: Sponsor
Organization: Akeso (Industry)
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Other
Other Study IDs: AK119-101
Record Dates: First submitted 2020-08-13; First posted 2020-08-18 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Coronavirus Disease 2019 (COVID-19)
Keywords: Anti-CD73; immunotherapy
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AK119 (Experimental): Single dose of AK119 is administered via intravenous infusion to healthy subjects.
  Interventions: Drug: AK119
- Placebo (Experimental): Single dose of placebo is administered via intravenous infusion to healthy subjects.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AK119 — Single dose of AK119 is administered via intravenous infusion to healthy subjects
  Arms: AK119
Drug: Placebo — Single dose of placebo is administered via intravenous infusion to healthy subjects
  Arms: Placebo

SUMMARY:
This is a first-in-human (FIH), Phase 1, single-center, randomized, double-blind, placebo-controlled, single ascending dose study to evaluate the safety, tolerability, PK and immunogenicity of AK119, a humanized monoclonal antibody targeting the CD73. The study will consist of 4 cohorts of healthy subjects. Eight subjects will be enrolled per cohort, randomized in a 3:1 ratio to receive a single dose of either the active drug AK119 (N=6) or matching placebo (N=2). Approximately 32 subjects (24 receiving active drug and 8 receiving placebo) will participate in this study.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet ALL the following inclusion criteria (as applicable) to be eligible for participation in this study:

* Adults between 18 and 55 years of age, inclusive, at screening.
* Must have a calculated body mass index (BMI, weight [kg]/height [m2]) within 18.0 to 30.0 kg/m2 (inclusive) at screening, and a total body weight ≥50 kg for men or ≥45 kg for women at screening and Day -1 before randomization.
* Must, in the opinion of the Investigator, be in good general health based upon medical history, physical examination (including vital signs), and 12-lead ECG; and clinical laboratory tests (up to 1 repeat permitted) must fall within the clinical laboratory"s reference normal ranges.

Exclusion Criteria:

Subjects who meet ANY of the following exclusion criteria will not be enrolled in this study

* Have a history of latent or active granulomatous infection, including histoplasmosis, candidiasis, or coccidioidomycosis prior to screening, or a history of any other infectious disease within 4 weeks prior to screening that, in the opinion of the Investigator, affects the subject"s ability to participate in the study.
* Have a history of multiple drug allergies or a known allergy or hypersensitivity to any biologic therapy at screening that is important in the opinion of the Investigator.
* Have a known allergy or reaction to any component of the AK119 formulation.
* Have any known malignancy or have a history of malignancy within the previous 5 years.
* Have a 12-lead ECG demonstrating QTcF interval > 450 msec for male subjects and >470 msec for female subjects at screening and Day -1 from average of 3 ECGs obtained after 5 minutes of supine rest.
* Blood pressure (BP) >150 mmHg (systolic) or > 95 mmHg (diastolic) at screening and Day -1, following at least 5 minutes of supine rest.
* Have had a live vaccination within 12 weeks prior to the study dosing or intend to have a live vaccination during the course of the study or have participated in a vaccine clinical study within 12 weeks prior to the study dosing.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2021-05-04 (Actual); Study Completion 2021-06-21 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent AEs | From signing of informed consent till end of study (approximately 64 days postdose)

SECONDARY OUTCOMES:
Maximum serum concentration (Cmax) of AK119 | From baseline till end of study (approximately 64 days postdose)
Area under the concentration-time curve (AUC) of serum concentration of AK119 | From baseline till end of study (approximately 64 days postdose)
Percentage of subjects who develop detectable anti-drug antibodies (ADAs) | From baseline till end of study (approximately 64 days postdose)

CONTACTS AND LOCATIONS:
Locations (1):
- Christchurch Clinical Studies Trust, Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343